CLINICAL TRIAL: NCT06110078
Title: Carbonic Anhydrase Inhibitors and Carbonation: A Novel Approach to Reduce Soda Consumption
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, C. William Heise MD, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003535
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Daily oral acetazolamide mouth rinse 10 ml
  Interventions: Drug: Acetazolamide
- Group 2 (Experimental): Twice daily oral acetazolamide mouth rinse 10 ml
  Interventions: Drug: Acetazolamide
- Group 3 (Placebo Comparator): Placebo mouth wash daily 10 ml
  Interventions: Drug: Acetazolamide
- Group 4 (Placebo Comparator): Twice daily placebo mouth wash 10 ml
  Interventions: Drug: Acetazolamide

INTERVENTIONS:
Drug: Acetazolamide — Oral rinse with acetazolamide (not taken orally)

SUMMARY:
Acetazolamide is a drug that is approved by the FDA for treating various conditions like epilepsy, altitude sickness, and glaucoma. Acetazolamide works by inhibiting an enzyme called carbonic anhydrase, which is important for many essential processes in our body. For example, carbonic anhydrase is needed to transport carbon dioxide in our blood which is essential for respiration.

One of the interesting effects of acetazolamide is that it reduces the taste of carbonation, making carbonated drinks like soda taste flat and or like soapy water. This effect has been noticed by hikers using the drug for mountain sickness treatment. It's believed that carbonic anhydrase inhibitors decrease the levels of carbonic acid in our mouths, which in turn reduces and changes the perception of carbonation taste.

It was hypothesized that this side effect of acetazolamide could be used to help people cut down on soda consumption. Since soda has been linked to health issues like obesity and type 2 diabetes, reducing its intake could be beneficial. In a case study, a person who took low-dose acetazolamide for six weeks experienced weight loss and found it easier to avoid carbonated drinks.

We are proposing a study to explore the effects of using acetazolamide as an oral rinse to decrease soda intake. The use of acetazolamide as an oral rinse has yet to be tested and is a possible way to decrease the taste of carbonation while also decreasing the side effects of the drug. Our plan is to use different doses of the rinse on participants and monitor their soda consumption and body mass index changes.

In summary, acetazolamide, a drug with various medical uses, could potentially help people reduce soda consumption by altering the taste of carbonation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Consumes on average ≥ 7 sodas per week
3. Healthy and without a history of significant neurological, liver, renal, cardiac or pulmonary disease.
4. No allergy to sulfa drugs or aspirin (contained in Alka Seltzer).
5. Ability to provide informed consent.

Exclusion Criteria:

Healthy adults, UA students, UA faculty and staff Exclusion Criteria:

1. Pregnant or lactating women.
2. Prisoners.
3. Refugees.
4. Cognitive impairment.
5. Chronic illness.
6. Allergy to sulfa drugs or aspirin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Soda intake | 3 weeks
  Total soda/carbonated beverage intake per week

SECONDARY OUTCOMES:
Weight | 3 weeks
  BMI/weight

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine Phoenix U of Arizona, Phoenix, Arizona, United States